CLINICAL TRIAL: NCT01135342
Title: Adding Sleep Intervention to Traditional Diet and Exercise Approach to Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine (Research), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SU-05062010-5883; 1R21HL092268-01A2 (NIH)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Sleep Initiation and Maintenance Disorders; Obesity
Keywords: Insomnia; Weight loss; Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Obesity; Weight Loss | interventions — Diet; Exercise; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet & Exercise plus Sleep Intervention (Experimental): Diet and exercise instruction to promote weight loss plus cognitive behavioral therapy for insomnia.
  Interventions: Behavioral: Diet and exercise; Behavioral: Cognitive Behavioral Therapy
- Diet & Exercise plus Passion and Balance (Sham Comparator): Diet and exercise instruction to promote weight loss plus sessions that are of general interest, but unrelated to diet, exercise, or sleep.
  Interventions: Behavioral: Diet and exercise; Behavioral: Passion and Balance

INTERVENTIONS:
Behavioral: Diet and exercise — Standardized instruction to eat less and exercise more to create an energy balance deficit to promote weight loss (16 classes)
Behavioral: Cognitive Behavioral Therapy — Standardized cognitive behavioral therapy for insomnia (8 classes)
  Arms: Diet & Exercise plus Sleep Intervention
Behavioral: Passion and Balance — Attention-match sessions of general interest, but unrelated to diet, exercise, or sleep (8 sessions)
  Arms: Diet & Exercise plus Passion and Balance

SUMMARY:
The goal is to determine if improved sleep will increase/enhance weight loss among overweight adults with insomnia.

DETAILED DESCRIPTION:
The major purpose of this study is to examine the effect of sleep quality and quantity on weight loss. The outcomes being studied are weight loss and improved sleep. The subjects being studied are those with body mass index 28-40kg/m2 who report sleeping less than 6.5 hours per day for 4 day per week or more for the past 6 months or longer and would likely benefit the most from the sleep intervention should it prove to be effective. We hope to learn if improved sleep habits among overweight adults with insomnia will help them to adhere to a diet and exercise program and increase their success with weight loss. Given the current world-wide obesity epidemic and the established difficulties many people have with weight control, any approaches that can be demonstrated to contribute to successful weight loss have direct public health significance.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both women and men
* Age: > or = 18 years
* Ethnicity and race: All ethnic and racial backgrounds welcome
* The following, which will be measured at the screening clinic visit:

  * Body Mass Index: 28-40 (kg/m-squared)
  * Chronic Short Sleep: total sleep time < 6.5 hours, greater than or equal to 4 days per week (determined by 1-week sleep log) for the past 6 months or longer (based on self-report).
  * Insomnia: sleep latency and/or wake after sleep onset > 30 minutes, greater than or equal to 4 days per week, insomnia severity index > 10, and complaint of at least one negative effect during waking hours (such as fatigue, sleepiness, impaired functioning, mood disturbance) attributed to sleep (as determined by self report).
  * Eligible sleep disorder: sleep apnea or upper airway resistance syndrome treated by positive airway therapy for > or = 3 months resulting in improved sleep.
  * Psychiatric disorders that are stable on SSRI, SNRI, or bupropion antidepressant for greater than or equal to 3 months if no anticipated changes in medications to occur during the trial if they are weight stable.
  * Planning to be available for clinic visits and for the 8 weeks of study participation
  * Ability and willingness to give written informed consent.

Exclusion Criteria:At screening:

* Sleep apnea (apnea-hypopnea index > 15/hr) determined by portable sleep diagnostic system Periodic limb movements during sleep (PLM with arousal index > 15/hr) determined by polysomnography.
* Any suspected sleep disorders identified by the Global Sleep Assessment Questionnaire, including circadian rhythm disorders (including shift work), parasomnias, narcolepsy, and restless leg.
* Self reported personal history of:
* DSM-IV Axis-I and Axis-II diagnoses (i.e. eating disorders, bi-polar disorder, schizophrenia and other psychotic disorders, substance-related disorders, personality disorders, poorly controlled major depression and anxiety disorders determined by SCID) except those allowed under Inclusions.
* Subjects currently receiving the following medications known to affect sleep(self report):

  * sedative hypnotics
  * sedative antidepressants
  * systemic steroids
  * anticonvulsants
  * histamine-1
  * receptor antagonists
  * narcotic analgesics
  * CNS stimulants
* Body Mass Index (BMI) greater than 40.
* Pregnant, Lactating, or <6 months post-partum.
* Inability to communicate effectively with study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight at 8 months | Baseline and 8 months
  Change was calculated as the value at 8 months minus the value at baseline.

SECONDARY OUTCOMES:
Change from baseline in scores of Insomnia Severity Index | Baseline and 8 months
  Change was calculated as the value at 8 months minus the value at baseline.
Change from baseline in scores of Insomnia Frequency Questionnaire | Baseline and 8 months
  Change was calculated as the value at 8 months minus the value at baseline.
Change from baseline in scores of Pittsburgh Sleep Quality Index | Baseline and 8 months
  Change was calculated as the value at 8 months minus the value at baseline.
Change from baseline in scores of Monk Social Rhythm Questionnaire | Baseline and 8 months
  Change was calculated as the value at 8 months minus the value at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study description and summary of results. — https://med.stanford.edu/nutrition/research/completed-studies/sleep-and-weight-loss.html